CLINICAL TRIAL: NCT06187519
Title: Cutaneous Uric Acid and Metabolite Monitor System (UR+AIMS) Lab Validation
Brief Title: UR+AIMS Gout Wearable Skin Uric Acid Monitor Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, John D. Fitzgerald, MD, PhD, Clin Prof, Clinical Chief, University of California, Los Angeles
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: UR+AIMS; R21DK132666 (NIH)
Record Dates: First submitted 2023-07-17; First posted 2024-01-02 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Gout
MeSH Terms: conditions — Gout | interventions — Transdermal Patch

STUDY DESIGN:
Intervention Model Description: 15 patients with gout [10 patients no recent urate-lowering therapy (ULT) and 5 patients on stable urate-lowering therapy (ULT)] will be invited to participate in a standardized meal at the UCLA Human Nutrition Center
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Uric Acid and Metabolite Monitor System (UR+AIMS) skin patch (Experimental): 15 patients with gout will be invited to participate in a standardized meal at the UCLA Human Nutrition Center and a 7-day community follow up for the measurement of uric acid (and other metabolites) using our Uric Acid and Metabolite Monitor System (UR+AIMS) skin patch.
  Interventions: Device: Uric Acid and Metabolite Monitor System (UR+AIMS) skin patch

INTERVENTIONS:
Device: Uric Acid and Metabolite Monitor System (UR+AIMS) skin patch — The intervention tested is the system (patch and mobile device/phone for reporting) that provides patients with better knowledge (test results) about the impact of their daily dietary choices on their uric acid levels.

SUMMARY:
15 patients with gout [10 patients no recent urate-lowering therapy (ULT) and 5 patients on stable urate-lowering therapy (ULT)] will be invited to participate in a standardized meal at the UCLA Human Nutrition Center and a 7-day community follow-up for the measurement of uric acid (and other metabolites) using our Uric Acid and Metabolite Monitor System (UR+AIMS) skin patch.

DETAILED DESCRIPTION:
First Visit at the UCLA Human Nutrition Center:

* Patients will sign the informed consent, then answer some study questionnaires.
* The Uric Acid and Metabolite Monitor System (UR+AIMS) skin patch and the study mobile device will be provided.
* Study nurse will start an IV for pre and post blood draws.
* Patients will be provided a standardized high-purine meal within 15 minutes. Pre-blood is drawn right before the patients eat the meal, then post-blood will be drawn every 15 minutes for the first hour after completion of the meal, then every 30 minutes for the next 3 hours (total of 4 hours).
* Then patients will be sent home with the skin patch and study mobile device.

Community 7-day observation period:

* Patients will be asked to apply a study patch each morning before their first meal of the day. The patch should be removed at the end of the day and put under water.
* The study device will monitor the patient's UA, glucose, heart rate, blood pressure, daily steps, and sleep. Patients will be asked to enter before and after meal uric acid levels and may be asked to take a picture of their meals using the study mobile device.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18 with diagnosis of gout (screening positive ACR/EULAR Gout Classification Criteria - see screening survey) and eGFR > 60 (within the last 12-months).
2. For the 10 patients with gout off urate-lowering therapy (ULT) [no Allopurinol, febuxostat, or probenecid prescription within the last 6-months] and serum urate (SU) > 7 mg/dL (within the last 12-months).
3. For the 5 patients with gout on urate-lowering therapy (ULT) [no dose change within the last 30 days].

Exclusion Criteria:

1. Contraindications to miosis, which include acute iritis, narrow-angle glaucoma
2. Known Hypersensitivity to pilocarpine hydrochloride
3. Pupillary block glaucoma (ophthalmic solution)
4. Subjects reporting any allergy to glue or latex or any allergy to food that will be provided in the study (sardines in extra virgin olive oil and Sprite).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2025-03-10 (Actual); Primary Completion 2025-06-18 (Actual); Study Completion 2025-09-03 (Actual)

PRIMARY OUTCOMES:
Evaluate tolerability and adherence of daily recorded patch wear time. | 3 years
  Daily recorded patch wear time as recorded by mobile phone app.
Recording of uric acid (and oxypurinol) measurements while wearing patch. | 3 years
  Recording of uric acid (and other metabolites e.g., uric acid, oxypurinol, ethanol) measurements while wearing patch recorded by patch Bluetooth to mobile phone.

CONTACTS AND LOCATIONS:
Overall Officials: John FitzGerald, MD, Principal Investigator — University of California, Los Angeles
Locations (1):
- UCLA, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Undecided